CLINICAL TRIAL: NCT05262946
Title: Somatosensory Restoration and Postural Control Improvement in People With Diabetic Peripheral Neuropathy Applying Sensorimotor Training: a Multicentric Randomized Controlled Trial
Brief Title: Sensorimotor Training for Adults With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DiabetesBalanceOne
Record Dates: First submitted 2022-01-31; First posted 2022-03-02 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Neuropathy; Somatosensory Disorders; Sensorimotor Gait Disorder
Keywords: gait; diabetes; sensorimotor training; peripheral neuropathy; somatosensory system; postural control; quality of life; fear of falling; Feldenkrais method
MeSH Terms: conditions — Peripheral Nervous System Diseases; Somatosensory Disorders; Gait Disorders, Neurologic; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 2 arms and single blinded randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: measurements and statistical analysis were made without knowing who participated in control or experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): control arm: usual care and foot care education.
  Interventions: Behavioral: foot care education; Combination Product: usual care
- experimental (Experimental): experimental arm: sensorimotor training, foot care education and usual care
  Interventions: Behavioral: sensorimotor training based on Feldenkrais method; Behavioral: foot care education; Combination Product: usual care

INTERVENTIONS:
Behavioral: sensorimotor training based on Feldenkrais method — 8 weeks of balance and sensorimotor training twice a week
  Arms: experimental
Behavioral: foot care education — Recommendations for preventing foot ulcers
Combination Product: usual care — drugs and diet usual care

SUMMARY:
Adults with diabetic peripheral neuropathy tend to fall more frequently than healthy population as a consequence of multiple sensorimotor and cognitive damages. In this protocol study, a randomized controlled trial is proposed using a sensorimotor intervention based on Feldenkrais method to improve somatosensory aspects and, therefore, postural control of participants.

DETAILED DESCRIPTION:
Among all the systems suffering damage due to hyperglucemia toxicity in diabetes, somatosensory system, composed by proprioception and skin sensory receptors has a key role since it is in charge of the faster body reaction when a postural control response is needed. Despite of it, few studies have focused on this issue. This randomized controlled trial proposed a safe and easy training adapted to adults and old people with diabetic peripheral neuropathy. Pressure, touch, proprioception and graphesthesia sensibility were measured, as well as functionality in daily basis, quality of life and fear of falling.

ELIGIBILITY:
Inclusion Criteria: having peripheral neuropathy and history of falls or risk factors for it. Current ulcer -

Exclusion Criteria: amputation and cognitive or mental issues

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Cumulative Somatosensory Impairment Index | 2 years
  It measures proprioception, pressure and vibration sensitivity and graphesthesia to sum up somatosensory function in lower legs. Iti is ranging from 0 to 8 being 8 the worst result

SECONDARY OUTCOMES:
Up and Go test | 2 years
  postural control test
Four Square Step test | 2 years
  ability walking in different directions
Tinetti- Performance-Oriented Mobility Assessment (POMA-T) | 2 years
  static and dynamic postural control
Falls Efficacy Scale | 2 years
  It measures the fear of falling, ranging from 0 to 64, being higher scores worst outcome results
SF-36 Health Survey questionnaire , 1.4 version. | 2 years
  Quality of life health-related questionnaire
Validated Spanish version of Short-Form Late-Life Function and Disability Instrument | 2 years
  It measures functional disabilities and frequency of daily life activities, ranging from 31 to 155 and being higher scores better outcome results.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA TERESA ANGULO CARRERA, DR, Study Director — UNIVERSIDAD COMPLUTENSE MADRID; NOEMI GONZALEZ PEREZ DE VILLAR, DR, Study Director — HOSPITAL UNIVERSITARIO DE LA PAZ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez-Mazuelas MJ, Gonzalez-Perez de Villar N, De Casas-Albendea S, Martinez-Gimeno L, Jimenez-Gonzalez S, Angulo-Carrere MT. Somatosensory and dynamic balance improvement in older adults with diabetic peripheral neuropathy through sensorimotor exercise: A multisite randomized controlled trial. J Bodyw Mov Ther. 2024 Oct;40:2062-2073. doi: 10.1016/j.jbmt.2024.10.041. Epub 2024 Oct 24. PMID 39593566